CLINICAL TRIAL: NCT07068724
Title: Chemical and Laser Desensitization Approaches for Managing Dentin Hypersensitivity After Non-Surgical Periodontal Therapy: A Randomized Clinical Trial
Brief Title: Management of Dentin Hypersensitivity in Patients With Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Ece AÇIKGÖZ ALPARSLAN, Assistant professor, Trakya University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-KAEK-06
Record Dates: First submitted 2025-04-10; First posted 2025-07-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-10

CONDITIONS: Dentin Hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — gluma desensitizer

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gluma applied group (No Intervention): Participants received Gluma Desensitizer (containing glutaraldehyde) applied to the sensitive teeth. Following isolation of the target teeth with cotton rolls, Gluma was applied using a microbrush in a rubbing motion for 30 seconds. The dentin surface was then air-dried until it lost its shine, followed by rinsing with water for 60 seconds.
- laser applied group (Experimental): Participants received Er,Cr:YSGG laser treatment (Water-Lase iPlusTM; Biolase® Technology Inc., Irvine, CA, USA). Laser parameters were set as follows: 2780 nm wavelength, 0.25 W power, 20 Hz frequency, 140 μs pulse duration, and 30 seconds exposure time. The MZ6 tip (660 μm diameter, 6 mm length, 1 mm spot size) was used in non-contact mode from a 1 mm distance, perpendicular to the dentin surface, with 0% water and 10% air spray. All laser applications followed international safety standards and protocols.
  Interventions: Device: Er,Cr:YSGG laser
- Combination applied group (Experimental): Participants in this group received both treatments: Gluma was applied using the same method as in Gluma, followed by Er,Cr:YSGG laser therapy using the same parameters and technique as in laser.
  Interventions: Combination Product: Gluma Desensitizer and ER:CR;YSGG laser combination

INTERVENTIONS:
Combination Product: Gluma Desensitizer and ER:CR;YSGG laser combination — Participants in this group received both treatments: Gluma was applied using the same method as in Gluma, followed by Er,Cr:YSGG laser therapy using the same parameters and technique as in laser.
  Arms: Combination applied group
Device: Er,Cr:YSGG laser — Participants received Er,Cr:YSGG laser treatment (Water-Lase iPlusTM; Biolase® Technology Inc., Irvine, CA, USA). Laser parameters were set as follows: 2780 nm wavelength, 0.25 W power, 20 Hz frequency, 140 μs pulse duration, and 30 seconds exposure time. The MZ6 tip (660 μm diameter, 6 mm length, 1 mm spot size) was used in non-contact mode from a 1 mm distance, perpendicular to the dentin surface, with 0% water and 10% air spray. All laser applications followed international safety standards and protocols.
  Arms: laser applied group

SUMMARY:
A total of 62 patients diagnosed with Stage III-IV periodontitis underwent non-surgical periodontal therapy. At 24 hours post-treatment, patients were recalled to the clinic for reassessment using air-stimulated Visual Analog Scale (VAS) and Schiff Cold Air Sensitivity Scale measurements. Two teeth per patient were randomly selected based on a VAS score greater than 4 and a Schiff score of 2 or 3. A total of 52 patients who met the inclusion criteria were included in the study. This study was designed as a randomized, parallel clinical trial. The 52 patients were randomly allocated into three treatment groups: Group 1 received the desensitizing agent Gluma, Group 2 underwent Er,Cr:YSGG laser treatment, and Group 3 received a combination of Gluma and Er,Cr:YSGG laser therapy. Desensitizing agent applications were performed according to the designated treatment protocols.To assess changes in dentin hypersensitivity over time, patients were recalled for follow-up evaluations at 1 week, 2 weeks, 1 month, 2 months and 6 months post-application. The 6-month follow-up of the study was completed with 48 patients (16 patients for each study group). At each follow-up visit, air-stimulated VAS and Schiff scale measurements were employed to quantify hypersensitivity levels.

ELIGIBILITY:
Inclusion Criteria:

* 1. No reported or clinically detected dentin hypersensitivity prior to the initiation of non-surgical periodontal therapy.

  2. Presence of at least five teeth with probing pocket depths (PPD) ≥6 mm. 3. Systemically healthy individuals with no history of systemic diseases that may interfere with periodontal outcomes.

  4. Absence of deep restorations or visible cracks in the teeth adjacent to those selected for hypersensitivity evaluation.

  5. No previous treatment for dentin hypersensitivity and no current use of desensitizing toothpaste or products.

  6. Clinical diagnosis of Stage III or IV periodontitis, involving periodontal support loss in more than 30% of teeth.

  7. A clinical attachment level (CAL) ≥5 mm and radiographic evidence of bone loss extending to the mid-root level.

  8. Age 18 years or older at the time of enrollment

Exclusion Criteria:

* 1. Use of antibiotics or analgesic medications at the time of screening or during the course of the study.

  2. Pregnancy or breastfeeding. 3. Receipt of periodontal therapy within the preceding 6 months. 4. Smoking history of 10 or more cigarettes per day. 5. Regular use of desensitizing toothpaste or other anti-hypersensitivity agents.

  6. Presence of parafunctional oral habits (e.g., bruxism, clenching). 7. Existence of non-carious cervical lesions such as erosion, attrition, or abrasion on study or adjacent teeth.

  8. High frequency of acidic dietary intake. 9. Inability to meet hypersensitivity perception thresholds following non-surgical periodontal therapy, defined as a Visual Analog Scale (VAS) score >4 and Schiff Cold Air Sensitivity Scale score of 2 or 3.

  10. Contraindications to the use of Er,Cr:YSGG laser therapy, including but not limited to: known allergies to local or topical anesthetics, presence of cardiac devices (e.g., pacemakers or implantable defibrillators), respiratory disease, bleeding disorders, or immunosuppressive conditions. In such cases, written clearance from a physician is required.

  11. Known or suspected allergy to any component of the Gluma Desensitizer, specifically hydroxymethyl methacrylate or glutaraldehyde.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2025-04-10 (Actual); Primary Completion 2025-10-10 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
Decrease in hypersensitivity rate | 6 months
  Combination of Gluma and Laser application can have an synergistic effect on hypersensitivity rate

CONTACTS AND LOCATIONS:
Locations (1):
- Trakya University, Edirne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated and/or analysed during the current study are not publicly available due to their sensitive and identifying nature, as well as the informed consent agreements made with participants but are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol